CLINICAL TRIAL: NCT05927909
Title: Validity and Reliability of the Turkish Version of the Low Back Activity Confidence Scale (Lobacs)
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Sezin Solum, MD; Physical Medicine & Rehabilitation Specialist Physician, Bursa City Hospital
Other Study IDs: 9999999992
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain, Mechanical; Symptoms and Signs
Keywords: low back pain; Turkish adaptation; validity; reliability; Low Back Activity Confidence Scale (Lobacs)
MeSH Terms: conditions — Low Back Pain; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Low Back Activity Confidence Scale (Lobacs) — Confidence Scale (LOBACS) is a self-report questionnaire designed to assess an individual's level of confidence in performing various physical activities involving the lower back region, to evaluate their perceived functional ability, and to assess the impact of low back pain on their daily life and functional performance.

SUMMARY:
Patients will be recruited from the Outpatient Department of Physical Medicine and Rehabilitation, Kestel State Hospital, who have been diagnosed with mechanical LBP for the past 3 weeks (physical examination, neurological examination, spinal radiography and laboratory tests and other causes of LBP were excluded) and who have agreed to participate in the study. Sociodemographic data of patients who gave written informed consent will be recorded to ensure anonymity. Although no consensus has been reached on the cross-cultural adaptation of the questionnaires into different languages, this study will use the guidelines for self-report measurement provided by Beaton et al. Following the formation of the expert committee, the scale will be translated and the pre-form back-translated. Comparisons will be made with the translated versions and the final version of the scale will be created by taking into account the opinions of the preliminary group of participants.

The reliability, test-retest reliability, face validity and content validity of the scale will be assessed by the expert committee. In order to assess the concurrent validity of this scale, all participants will also complete the 'Oswestry Low Back Pain Disability Questionnaire' and the 'Quebec Low Back Pain Disability Questionnaire', which have been previously validated and reliable in Turkish.

The Oswestry Low Back Pain Disability Questionnaire consists of 10 items that assess activities of daily living. These are pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, travelling and degree of change in pain. Each item has 6 options ranging from 0 to 5 points (12). The Quebec Low Back Pain Disability Questionnaire consists of 20 items assessing activities of daily living. Each item has 6 options ranging from 0-5 points.

The aim of this study was to evaluate the validity and reliability and the Turkish version of the Low Back Activity Confidence Scale (Lobacs).

DETAILED DESCRIPTION:
Patients will be recruited from the Outpatient Department of Physical Medicine and Rehabilitation, Kestel State Hospital, who have been diagnosed with mechanical LBP for the past 3 weeks (physical examination, neurological examination, spinal radiography and laboratory tests and other causes of LBP were excluded) and who have agreed to participate in the study. Sociodemographic data of patients who gave written informed consent will be recorded to ensure anonymity. Although no consensus has been reached on the cross-cultural adaptation of the questionnaires into different languages, this study will use the guidelines for self-report measurement provided by Beaton et al. Following the formation of the expert committee, the scale will be translated and the pre-form back-translated. Comparisons will be made with the translated versions and the final version of the scale will be created by taking into account the opinions of the preliminary group of participants.

The reliability, test-retest reliability, face validity and content validity of the scale will be assessed by the expert committee. In order to assess the concurrent validity of this scale, all participants will also complete the 'Oswestry Low Back Pain Disability Questionnaire' and the 'Quebec Low Back Pain Disability Questionnaire', which have been previously validated and reliable in Turkish.

The aim of this study was to evaluate the validity and reliability and the Turkish version of the Low Back Activity Confidence Scale (Lobacs).

ELIGIBILITY:
Inclusion Criteria:

* Presence of mechanical low back pain for 3 weeks or more.

Exclusion Criteria:

* Duration of pain is less than 3 weeks,
* Evidence of non-mechanical causes of low back pain on imaging or laboratory tests.
* Inflammatory diseases.
* History of major surgery in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Outpatient Department of Physical Medicine and Rehabilitation, Kestel State Hospital, who have been diagnosed with mechanical LBP for the past 3 weeks (physical examination, neurological examination, spinal radiography and laboratory tests and other causes of LBP were excluded) and who have agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Low Back Activity Confidence Scale (Lobacs) | baseline
  The Low Back Activity Confidence Scale (LOBACS) is a self-report questionnaire comprising 15 items and three subscales: Functional Self-efficacy (FnSE), Self-regulatory Self-efficacy, and Exercise Self-efficacy (ExSE). Its purpose is to evaluate an individual's perceived functional ability and the impact of low back pain on their daily life and functional performance. The questionnaire employs an 11-point Likert scale, ranging from 0% (no confidence) to 100% (complete confidence), with 10% increments for each point. Scores can be calculated globally (e.g., average score of all items) or for specific domains (e.g., average score of items 1-7 for FnSE subscale). The total score can range from 0 to 100, where higher scores indicate greater self-efficacy.
The Oswestry Back Pain Disability Questionnaire | baseline
  The Oswestry Back Pain Disability Questionnaire comprises 10 items that inquire about various daily activities, including pain intensity, self-care, lifting, walking, sitting, standing, sleeping, social life, traveling, and the extent of pain-related changes. Each item presents six response options, scored on a scale of 0 to 5 points.
The Quebec back pain disability scale (QBPDS) | baseline
  The Quebec Back Pain Disability Scale consists of 20 daily activities that can be categorised into 6 types of activities: Sitting/standing, Walking, Moving, Bending, Bed/resting, Handling large/heavy objects. For each activity there are 6 response scores on a Likert scale from 0-5 (0 = no effort, 5 = unable). If the person feels really bad, they give it a score of 5. If they feel good with no problems, they give it a score of 0.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Salbaş, MD, Study Director — Balikesir University
Locations (1):
- Bursa Kestel State Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yamada KA, Lewthwaite R, Popovich JM Jr, Beneck GJ, Kulig K; Physical Therapy Clinical Research Network. The Low Back Activity Confidence Scale (LoBACS): preliminary validity and reliability. Phys Ther. 2011 Nov;91(11):1592-603. doi: 10.2522/ptj.20100135. Epub 2011 Aug 18. PMID 21852520
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Chung KC, Pillsbury MS, Walters MR, Hayward RA. Reliability and validity testing of the Michigan Hand Outcomes Questionnaire. J Hand Surg Am. 1998 Jul;23(4):575-87. doi: 10.1016/S0363-5023(98)80042-7. PMID 9708370
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Melikoglu MA, Kocabas H, Sezer I, Bilgilisoy M, Tuncer T. Validation of the Turkish version of the Quebec back pain disability scale for patients with low back pain. Spine (Phila Pa 1976). 2009 Mar 15;34(6):E219-24. doi: 10.1097/BRS.0b013e3181971e2d. PMID 19282728
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN checklist for assessing the methodological quality of studies on measurement properties of health status measurement instruments: an international Delphi study. Qual Life Res. 2010 May;19(4):539-49. doi: 10.1007/s11136-010-9606-8. Epub 2010 Feb 19. PMID 20169472